CLINICAL TRIAL: NCT04936009
Title: Noninvasive Brain Stimulation to Treat Core Social Deficits in Autism Spectrum Disorder
Brief Title: Transcranial Magnetic Stimulation (TMS) Study for Adults With Autism Spectrum Disorder (ASD)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2000030576; Proposal No. AR200174 (Other Grant/Funding Number: Department of Defense)
Record Dates: First submitted 2021-06-13; First posted 2021-06-23 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Autism Spectrum Disorder
Keywords: Transcranial Magnetic Stimulation
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: Participants will receive both active and sham TMS in a randomized crossover assignment involving two study sessions.
Who Masked: Participant
Masking Description: Participants will not know whether they are receiving active or sham TMS until both sessions have been completed.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transcranial Magnetic Stimulation - real (Active Comparator): Participants will receive active TMS during their study visit
  Interventions: Behavioral: Transcranial Magnetic Stimulation (TMS)
- Transcranial Magnetic Stimulation - sham (Placebo Comparator): Participants will receive sham stimulation during their study visit simulating TMS
  Interventions: Behavioral: Transcranial Magnetic Stimulation (TMS)

INTERVENTIONS:
Behavioral: Transcranial Magnetic Stimulation (TMS) — Subjects will receive both active and sham TMS in a randomized crossover assignment involving two study sessions

SUMMARY:
This is a randomized interventional study designed to evaluate the effects of repetitive Transcranial Magnetic Stimulation (rTMS) on neural and behavioral facets of social cognition in adults with autism spectrum disorder (ASD).

DETAILED DESCRIPTION:
The primary objective of this study is to determine whether rTMS increases the brain response to faces in a population of adults with ASD. This study will assess critical aspects of social cognition using the electroencephalogram (EEG), event-related potentials (ERPS), and eye-tracking (ET) prior to and following a single rTMS session (or Sham) to provide preliminary insight into the potential of rTMS as a tool to modify social brain function in this population.

Participant visits will include a baseline assessment of neuropsychological, cognitive and behavioral function, and a pre and post TMS session with EEG (electroencephalogram) and eye-tracking to measure neural and visual attentional social response. Two study visits will be scheduled for each participant lasting approximately 4-5hrs total.

ELIGIBILITY:
Inclusion Criteria:

* Individuals between the ages of 18 and 40 years old with typical development or with a diagnosis of autism spectrum disorder.
* Individuals able to participate in an EEG and eye-tracking experiment.

Exclusion Criteria:

* Participants reporting significant head trauma or serious brain illness.
* Participants with major psychiatric illness that would preclude completion of study measures.
* Participants with a history of serious medical illness, stroke, seizures, epileptiform EEG abnormalities, or family history of seizures.
* Participants taking prescription medications that may affect cognitive processes under study.
* Participants who have taken alcohol or recreational drugs within the preceding 24 hours.
* Females of known/suspected pregnancy or who test positive on a pregnancy test.
* Participants with a history of metalworking or injury by shrapnel or metallic objects are also excluded.
* Participants with a history of prior TMS therapy or use of an investigational drug within 12 weeks of visit.
* Participants with an IQ (intelligence quotient) below 80.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-03-17 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
right hemisphere N170 latency | Measures will be recorded during the EEG/ET sessions of participant visits for an expected 1-2 hours
  EEG brain response to faces as measured by the N170 component in milliseconds
proportion of visual attention to the eye region of the face | Measures will be recorded during the EEG/ET sessions of participant visits for an expected 1-2 hours
  visual attention to the eye region of the face as measured by eye tracking in seconds

CONTACTS AND LOCATIONS:
Overall Officials: James McPartland, PhD, Principal Investigator — Yale University
Locations (1):
- Yale University Child Study Center, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rossi S, Hallett M, Rossini PM, Pascual-Leone A; Safety of TMS Consensus Group. Safety, ethical considerations, and application guidelines for the use of transcranial magnetic stimulation in clinical practice and research. Clin Neurophysiol. 2009 Dec;120(12):2008-2039. doi: 10.1016/j.clinph.2009.08.016. Epub 2009 Oct 14. PMID 19833552
- [Background] Huang YZ, Edwards MJ, Rounis E, Bhatia KP, Rothwell JC. Theta burst stimulation of the human motor cortex. Neuron. 2005 Jan 20;45(2):201-6. doi: 10.1016/j.neuron.2004.12.033. PMID 15664172
- [Background] Allison T, Puce A, McCarthy G. Social perception from visual cues: role of the STS region. Trends Cogn Sci. 2000 Jul;4(7):267-278. doi: 10.1016/s1364-6613(00)01501-1. PMID 10859571
- [Background] McPartland J, Dawson G, Webb SJ, Panagiotides H, Carver LJ. Event-related brain potentials reveal anomalies in temporal processing of faces in autism spectrum disorder. J Child Psychol Psychiatry. 2004 Oct;45(7):1235-45. doi: 10.1111/j.1469-7610.2004.00318.x. PMID 15335344
- [Background] Dawson G, Toth K, Abbott R, Osterling J, Munson J, Estes A, Liaw J. Early social attention impairments in autism: social orienting, joint attention, and attention to distress. Dev Psychol. 2004 Mar;40(2):271-83. doi: 10.1037/0012-1649.40.2.271. PMID 14979766
- [Background] Oberman LM, Rotenberg A, Pascual-Leone A. Use of transcranial magnetic stimulation in autism spectrum disorders. J Autism Dev Disord. 2015 Feb;45(2):524-36. doi: 10.1007/s10803-013-1960-2. PMID 24127165
- [Background] Abujadi C, Croarkin PE, Bellini BB, Brentani H, Marcolin MA. Intermittent theta-burst transcranial magnetic stimulation for autism spectrum disorder: an open-label pilot study. Braz J Psychiatry. 2018 Jul-Sep;40(3):309-311. doi: 10.1590/1516-4446-2017-2279. Epub 2017 Dec 11. PMID 29236921
- [Background] Ni HC, Hung J, Wu CT, Wu YY, Chang CJ, Chen RS, Huang YZ. The Impact of Single Session Intermittent Theta-Burst Stimulation over the Dorsolateral Prefrontal Cortex and Posterior Superior Temporal Sulcus on Adults with Autism Spectrum Disorder. Front Neurosci. 2017 May 9;11:255. doi: 10.3389/fnins.2017.00255. eCollection 2017. PMID 28536500